CLINICAL TRIAL: NCT04206358
Title: An Open Phase Ib Clinical Study to Evaluate OrienX010 in Combination With JS001 in the Treatment of Stage IV (M1c) Liver Metastasis From Melanoma
Brief Title: Study to Evaluate OrienX010 in Combination With JS001 in the Treatment of Stage IV (M1c) Liver Metastasis From Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of department of renal cancer and melanoma, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OrienX010-II-11
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Melanoma
Keywords: melanoma, Liver Metastasis
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): The Recombinant Human GM-CSF Herpes Simplex Virus Injection (OrienX010) in Combination with Recombinant Human Anti-PD1 Monoclonal Antibody Injection (JS001), Once every 2 weeks
  Interventions: Biological: OrienX010 combination with JS001

INTERVENTIONS:
Biological: OrienX010 combination with JS001 — OrienX010 Produced by Oriengene Biotechnology Co., Ltd. Strength: 1.0 mL/vial. Label claim: Titer 8.0 × 10^7Pfu/mL, NMT 1 × 10 particles11VP/mL.
  JS001 Produced by Junshi Biosciences Co., Ltd. Strength: 240 mg/6 mL/vial; Sterile water injection dosage form; Expiry date: 24 months; Date of manufacture: Based on the date of manufacture indicated in the product package.
  Other Names: Recombinant Human GM-CSF Herpes Simplex Virus Injection combination with Recombinant Human Anti-PD-1 Monoclonal Antibody Injection

SUMMARY:
This study is an open-label, Phase Ib clinical study to evaluate Evaluate the Recombinant Human GM-CSF Herpes Simplex Virus Injection (OrienX010) in Combination with Recombinant Human Anti-PD1 Monoclonal Antibody Injection (JS001) in the Treatment of Stage IV (M1c) Liver Metastasis from Melanoma.

This study is planned to enroll approximately 30 patients with Stage IV (M1c) Liver Metastasis from Melanoma who meet protocol requirements. This study is a single-arm clinical trial.

All participator will be given OrienX010 in combination with JS001. JS001 injection: 3 mg/kg, IV infusion: Once every 2 weeks ; OrienX010: Maximum injection volume 8 × 10^8 pfu, intratumoral injection: Once every 2 weeks. Treatment will be continuous and extend from first dose of study medication until to complete response, clinical related progression disease (PDr), intolerable AE, or withdrew informed consent or meet other criteria of discontinuation.

For patients who have stopped the study treatment and no disease progression, follow-up visits will take place every 3 months after the end of treatment visit until the occurrence of disease progression. If disease progression occurred, the investigator will collect the anticancer treatment information and survival of individuals until 80% death event.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain the current IRB approved informed consent with written from potential patients before the any screening activities or procedures.
2. Male or female, ≥ 18 years of age.
3. Patients with definite diagnosis of IV (M1c) Liver metastasis from melanoma based on histology and/or cytology.Patients who lack existing therapies or fail or relapse with existing therapies.
4. Patients with at least one injectable lesion on the liver (long diameter ≥ 10 mm and < 100 mm).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Expected Survival> 4 months;
7. The patients has good function in each organ, and the following conditions are required at screening according to the laboratory reference range:

   White blood cell count ≥ 3.0 × 109/L; Absolute neutrophil value ≥ 1.5 × 109/L; Platelet count ≥ 100 × 109/L; Hemoglobin ≥ 90 g/L; Serum albumin ≥ 2.5 g/dL; Liver function tests: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × ULN; Renal function tests: Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min at 24 hours (Cockcroft and Gault formula); International normalized ratio (INR) ≤ 1.5, and activated partial thromboplastin time (APTT) or partial prothrombin time (PTT) ≤ 1.5 × ULN;
8. Child-Pugh Grade A;
9. Patients receiving treatment for the first time in this study from the date of the last previous anti-tumor treatment date interval more than 28 days, and Patients have recovered from adverse events as a result of prior anti-tumor therapy to less than or equal to Grade 1, according to Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) (Except alopecia).
10. Female patients with childbearing potential (including premature menopause, menopausal < 2 years and non-surgical sterilization), male patients, and partners of male patients must agree to use effective contraception during the study: Surgical sterilization, oral contraceptives, intrauterine devices, sexual abstinence or barrier contraceptive combination spermicides; All patients must continue contraception for 6 months after the last treatment

Exclusion Criteria:

1. Patients previously treated with T-VEC or similar.
2. Patients previously treated with anti-PD-1, anti-PD-L1, anti-PD-L2.
3. Patients with negative anti-herpes simplex virus type I (HSV-1) antibodies IgG and IgM.
4. The patient's lesion does not meet the requirement of the intratumoral injection volume or is not suitable for intratumoral injection.
5. Received anti-herpes simplex virus therapy (such as aciclovir, ganciclovir, valaciclovir, and arabinoside) within 4 weeks prior to the first dose of study treatment.
6. Received another anti-tumor monoclonal antibody (mAb) within 4 weeks prior to the first dose of study treatment or hasn't recover (≤ Grade 1) from adverse events due to prior therapy (occurring earlier than 4 weeks;
7. Patients with a history of other (including unknown primary) malignancies within 5 years prior to the first dose of trial treatment. Note: Except for fully treated stage 1 or 2 basal/squamous cell carcinoma of the skin, superficial bladder cancer, or in situ cancer that is treated with potentially curative therapy.
8. Patients with known hypersensitivity to the study drug, its active ingredient, excipients.
9. Patient with HBsAg positive and HBV DNA copies > 1×10^3copies/mL.
10. Patients with positive hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies.
11. Patients with any unstable systemic disease, including but not limited to: Serious infection, uncontrolled diabetes mellitus, unstable angina, cerebrovascular accident or transient cerebral ischemia, myocardial infarction, congestive heart failure, and serious arrhythmia liver, kidney, or metabolic disease requiring medical treatment.
12. patients with active CNS metastases. patients may participate in the study if their CNS is adequately treated and their neurological symptoms recover to levels less than or equal to CTCAE1 for at least 2 weeks before enrollment, with the exception of residual signs or symptoms associated with CNS therapy . In addition, patients must be those who do not use corticosteroids or who take stable doses of ≤ 10 mg prednisone/day (or equivalent dose) or who decrease to ≤ 10 mg prednisone/day.
13. Patients with meningeal carcinomatosis.
14. Patients with autoimmune disease.
15. The disease (e.g., mental illness, etc.) or condition (e.g., alcoholism or drug abuse, etc.) of the patient may increase the patient's risk of receiving trial medication or affect the patient's compliance with the study requirements, or may confuse the study results.
16. Within 30 days of screening, the patient had received any other study product or had participated in another intervention clinical trial.
17. Pregnant or lactating women, or women who are prepared to become pregnant or lactating during the study; Men or women who are unwilling to use effective contraception.
18. Other situations that the investigators think are not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-02-27 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of enrolling until subjects disease progressive, an average of 16 weeks
  Progression-free survival (PFS), defined as the first documentation of objective disease progression, according to Response Evaluation Criteria in Solid Tumors (RECIST v.1.1)
ORR | From date of enrolling until the date of all patients disease progression , an average of 20 months.
  Objective Response Rate (ORR), defined as complete or partial tumor response, according to RECIST v.1.1 criteria

SECONDARY OUTCOMES:
OS | Approximately 3 years
  Overall survival defined as the time from randomization to death from any cause
Quality of life assessment | every 8 weeks, up to the date of 28 days after stopping treatment, an average of 24 weeks
  Use EORTC QLQ-C30 to assess quality of life. The EORTC(European Organization for Research and Treatment of Cancer) QLQ-C30 (Quality of Life Questionnaire C30), is a cancer-specific quality of life instrument applicable to a broad range of cancer patients.
  QLQ-C30 contain 15 domain, The standard score for each domain from 0-100. higher scores mean a worse outcome.
Incidence of SAE and AE | From date of enrolling to 90 days after stopping treatment, an average of 20 months
  Number of AE (adverse events) and SAE (serious adverse events) occurrences， Number of participants with treatment-related SAE and AE that assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No